CLINICAL TRIAL: NCT01871324
Title: The Efficacy of Group Therapy in Ultra-Orthodox Jewish Young Men Diagnosed With Type One Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: technical issues
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ofri Mosenzon, Head of Diabetes Research Unit, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0560-12-HMO-CTIL
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Behavioral Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — group therapy

SUMMARY:
The purpose of this study is to compare the influence of an intervention program especially designed to young ultra orthodox men that were diagnosed with diabetes type one.

ELIGIBILITY:
Inclusion Criteria:

* Young Ultra-Orthodox men diagnosed with diabetes type one.

Exclusion Criteria:

* Psychiatric illness .

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Estimated); Primary Completion 2015-09 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
the efficacy will be evaluated using Diabetes Quality of Life questionnaire before and after the program. | three months

SECONDARY OUTCOMES:
the efficacy will be evaluated using behavioral changes related to diabetes questionnaire before and after the program. | three months

OTHER OUTCOMES:
the efficacy will be evaluated using HbA1c values, glucose levels before and after the program | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel